CLINICAL TRIAL: NCT03847207
Title: A Three-Part Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Ascending Subcutaneous Doses of HTL0030310 in Healthy Subjects
Brief Title: A Study in Healthy Subjects to Assess the Safety, Tolerability, PK and PD of HTL0030310
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nxera Pharma UK Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: HTL0030310-101; 2018-003169-33 (EudraCT Number); QSC200729 (Other: Quotient Sciences)
Record Dates: First submitted 2019-01-18; First posted 2019-02-20 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Healthy
Keywords: First in Human; Single Ascending Dose
MeSH Terms: interventions — pasireotide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1 Single Ascending Dose (Experimental): Eight subjects in up to 8 cohorts will be dosed. A single subcutaneous injection of HTL0030310 or placebo will be administered. In each cohort, 6 subjects will receive HTL0030310 and 2 subjects will receive placebo.
  Interventions: Drug: HTL0030310; Drug: Placebo
- Part 2 Pasireotide PD Assessment (Experimental): Sixteen subjects in 2 cohorts (8 subjects per cohort) will be dosed on 4 occasions. Within each cohort, 4 subjects will be randomised to active dosing with CRH with desmopressin, GHRH and OGTT challenge and 4 subjects will be randomised to placebo dosing with CRH with desmopressin, GHRH and OGTT challenge.
  Interventions: Drug: Pasireotide; Drug: Placebo
- Part 3 Proof of Pharmacological Effect (Experimental): Up to 80 subjects in 4 cohorts (up to 20 subjects per cohort) will be dosed in up to 3 study periods. In each period, subjects will receive active drug or placebo with GHRH, OGTT and CRH with desmopressin (optional).
  Interventions: Drug: HTL0030310; Drug: Placebo

INTERVENTIONS:
Drug: HTL0030310 — Solution for Subcutaneous injection
  Arms: Part 1 Single Ascending Dose; Part 3 Proof of Pharmacological Effect
Drug: Pasireotide — Pasireotide 600 μg for subcutaneous injection
  Arms: Part 2 Pasireotide PD Assessment
Drug: Placebo — Matching placebo Solution

SUMMARY:
A Phase 1, first in human, three-part, single centre study to assess the safety, tolerability, PK and PD of single ascending subcutaneous doses of HTL0030310 in healthy subjects

DETAILED DESCRIPTION:
This is a first in human, three part study with the objective to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of single ascending subcutaneous doses of HTL0030310 in healthy subjects. Part 1 is a double-blind, placebo-controlled, randomised study assessing single ascending doses of HTL0030310. Part 2 is a site-blind (sponsor unblinded), placebo-controlled, part-randomised, fixed-sequence, single-dose, 4-period study assessing the PD of a positive control, pasireotide, following administration of challenge agents. Part 3 is a double-blind, placebo-controlled, part-randomised, fixed-sequence, single-dose, HTL0030310 proof of pharmacological effect study, where PD effects of HTL0030310 will be investigated following administration of challenge agents. The challenge agents administered in this study will be: oral glucose tolerance test (OGTT), Growth hormone-releasing hormone (GHRH), and corticotrophin releasing hormone (CRH) combined with desmopressin.

ELIGIBILITY:
Inclusion Criteria

1. Healthy males or healthy a woman is considered of childbearing potentiaL (WONCBP); a WONCBP unless she is permanently sterile (hysterectomy, bilateral salpingectomy and bilateral oophorectomy) or is postmenopausal (had no menses for 12 months without an alternative medical cause and a serum follicle-stimulating hormone [FSH] concentration ≥40 IU/L).
2. Age 18 to 50 years of age
3. A BMI of 20.0 to 30.0 kg/m2, with a minimum weight of 45 kg
4. Must be willing and able to communicate and participate in the whole study
5. Must provide written informed consent
6. Must agree to adhere to the contraception requirements defined in the protocol (Section 9.4)

Exclusion Criteria

1. Subjects who have received any IMP in a clinical research study within the previous 3 months of screening
2. Subjects who are study site employees, or immediate family members of a study site or sponsor employee
3. Subjects who have previously been enrolled in this study. Subjects who have taken part in Part 1/Part 2 are not permitted to take part in Part 2/Part 3
4. History of any drug or alcohol abuse in the past 2 years
5. Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 Units = 125 mL glass of wine, depending on type)
6. Current smokers and those who have smoked within the last 12 months. A breath carbon monoxide reading of greater than 10 ppm at screening and admission
7. Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months
8. Females of childbearing potential. A woman is considered of childbearing potential unless she is permanently sterile (hysterectomy, bilateral salpingectomy and bilateral oophorectomy) or is postmenopausal (had no menses for 12 months without an alternative medical cause and a serum FSH concentration ≥40 IU/L). All female subjects must have a negative urine pregnancy test
9. Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator at screening
10. Subjects with vital signs outside the normal range for healthy volunteers (HR < 50 or >90 bpm; Systolic BP > 140 mmHg; Diastolic BP > 90 mmHg)
11. Clinically significant abnormal biochemistry, haematology, coagulation or urinalysis as judged by the investigator (laboratory parameters are listed in Appendix 1 of the protocol)
12. Fasting blood glucose at screening above the upper limit of normal (3.9 to 5.8 mM)
13. HbA1c at screening above the upper limit of normal (>6%)
14. Abnormal renal function - defined as creatinine clearance < 70mL/min using the Cockcroft-Gault equation at screening
15. Abnormal hepatic function - defined as ALT, AST and total bilirubin > 1.5 x upper limit of normal at screening
16. Positive drugs of abuse test result (drugs of abuse tests are listed in Appendix 1 of the protocol)
17. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
18. History of clinically significant cardiovascular, renal, hepatic, chronic respiratory or GI disease, neurological or psychiatric disorder, as judged by the investigator
19. Family history of long QT syndrome or sudden cardiac death in a young adult where a cause of arrhythmia cannot be excluded
20. QTcF at screening >450 msec in males or >470 msec in females
21. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients, including glucose/fructose intolerance for the standard OGTT
22. Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hayfever is allowed unless it is active
23. Donation or loss of greater than 400 mL of blood within the previous 3 months
24. Subjects who are taking, or have taken, any prescribed or over-the-counter drug (other than up to 4 g per day paracetamol) or herbal remedies (including St. John's Wort) in the 21 days before IMP administration (See Section 11.4 of protocol). Exceptions may apply on a case by case basis, if considered not to interfere with the objectives of the study, as agreed by the PI and sponsor's medical monitor
25. Subjects with tattoos or scars on the abdomen which may interfere with injection site assessments or pharmacodynamic measurements, as determined by the PI or delegate at screening
26. Failure to satisfy the investigator of fitness to participate for any other reason Exclusion criteria 11, 16, 22, 24 and 26 from the list above will be re-assessed at admission/pre-dose.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of treatment related adverse events (as determined by abnormal clinical laboratory tests, vitals signs, ECG parameters, Holter ECG parameters and injection site reactions) | Admission up to 8 days post dose
  Safety and Tolerability
Part 2 and Part 3 Area under the effect time curve (EAUC) 1) for insulin, glucose, glucagon, GLP1, C-peptide and GIP level 2) for GH 3) ACTH and cortisol | Predose up to 4 hours post dose
  Pharmacodynamics
Part 2 and Part 3 Maximum observed effect (EMax) 1) for insulin, glucose, glucagon, GLP1, C-peptide and GIP level 2) for GH 3) ACTH and cortisol | Predose up to 4 hours post dose
  Pharmacodynamics
Part 2 and Part 3 Time to reach Maximum observed effect (TEMax) 1) for insulin, glucose, glucagon, GLP1, C-peptide and GIP level 2) for GH 3) ACTH and cortisol | Predose up to 4 hours post dose
  Pharmacodynamics

SECONDARY OUTCOMES:
Part 1 Maximum observed plasma concentration (Cmax) of single subcutaneous doses of HTL0030310 | Pre dose to 144 hours post dose
  Pharmacokinetics
Part 1 Time to reach Maximum observed plasma concentration (Tmax) of single subcutaneous doses of HTL0030310 | Pre dose to 144 hours post dose
  Pharmacokinetics
Part 1 Area under the curve (AUC) of single subcutaneous doses of HTL0030310 | Pre dose to 144 hours post dose
  Pharmacokinetics
Part 2 Maximum observed plasma concentration (Cmax) of single subcutaneous doses of pasireotide | Predose to 24 hours postdose
  Pharmacokinetics
Part 2 Time to reach Maximum observed plasma concentration (Tmax) of single subcutaneous doses of pasireotide | Predose to 24 hours postdose
  Pharmacokinetics
Part 2 Area under the curve (AUC) of single subcutaneous doses of pasireotide | Predose to 24 hours postdose
  Pharmacokinetics
Part 3: Number of treatment related adverse events (as determined by abnormal clinical laboratory tests, vitals signs, ECG parameters and injection site reactions) | Admission up to 8 to 10 days post final dose
  Safety and Tolerability
Part 3 Maximum observed plasma concentration (Cmax) of single subcutaneous doses of HTL0030310 | Predose to 96 hours postdose
  Pharmacokinetics
Part 3 Time to reach Maximum observed plasma concentration (Tmax) of single subcutaneous doses of HTL0030310 | Predose to 96 hours postdose
  Pharmacokinetics
Part 3 Area under the curve (AUC) of single subcutaneous doses of HTL0030310 | Predose to 96 hours postdose
  Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Philip Evans, MBChB, Principal Investigator — Quotient Sciences
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No